CLINICAL TRIAL: NCT03174639
Title: High Myopia Macular Hole and Retinal Detachment Accepted Internal Limiting Membrane Flip Packing and Free Flap Was the Internal Limiting Membrane (ILM Flap Was Double)
Brief Title: High Myopia Macular Hole and Retinal Detachment Treated With Double ILM Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201512113RINA
Record Dates: First submitted 2017-05-23; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: High Myopia; Macular Holes; Retinal Detachment
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inverted and free ILM insertion (Experimental): Both inverted and free ILM flaps were inserted into the macular hole
  Interventions: Procedure: Inverted and free ILM insertion

INTERVENTIONS:
Procedure: Inverted and free ILM insertion — ILM was peeled and the ILM flap was inverted and inserted into the macular hole, followed by insertion of free ILM flap.

SUMMARY:
From July 2015 to December 2015, clinical record of 8 consecutive cases of macular hole with retinal detachment in high myopia treated with combined inverted and free ILM flap insertion into the hole were retrospectively reviewed. The anatomical and function outcomes were assessed.

DETAILED DESCRIPTION:
From July 2015 to December 2015, clinical record of 8 consecutive cases of macular hole with retinal detachment in high myopia treated with combined inverted and free ILM flap insertion into the hole were retrospectively reviewed. The anatomical and function outcomes were assessed. Patients with a history of trauma or concurrent peripheral breaks were excluded. The anatomical and function outcomes, including the status of the macular hole and retina were assessed.The study was approved by the ethnic committee and research board.

ELIGIBILITY:
Inclusion Criteria:

* Macular hole with retinal detachment in high myopia

Exclusion Criteria:

* History of trauma, peripheral retinal breaks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Closure of macular hole | 3 months
  Closure of macular hole demonstrated by optical coherence tomography

SECONDARY OUTCOMES:
Retinal reattachment | 3 months
  Retinal reattachment observed by fundoscopy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen SN, Yang CM. Double Internal Limiting Membrane Insertion for Macular Hole-Associated Retinal Detachment. J Ophthalmol. 2017;2017:3236516. doi: 10.1155/2017/3236516. Epub 2017 Jul 30. PMID 28845304